CLINICAL TRIAL: NCT04366024
Title: A Novel Nomogram to Predict Severity of COVID-19
Status: Completed | Type: Observational
Sponsor: Xinqiao Hospital of Chongqing (Other)
Responsible Party: Principal Investigator, Jianguo Sun, Deputy Director,Head of Oncology department, Principal Investigator, Clinical Professor, Xinqiao Hospital of Chongqing
Other Study IDs: XQonc-016
Record Dates: First submitted 2020-04-21; First posted 2020-04-28 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: COVID-19 Disease; Nomogram Model

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observed group: COVID-19 disease patients who were detected by RT-PCR and CT imaging.
  Interventions: Other: other

INTERVENTIONS:
Other: other — clinical diagnosis

SUMMARY:
Investigators use clinical data from a large sample of COVID-19 disease patients to screen out biomarkers associated with disease severity. Then, a novel nomogram model will be established to predict covid-19 disease severity, which could provide important assistance and supplement for clinical work. In the case of extremely shortage of front-line medical resources, patients with potential severe diseases will be timely treated with the help of the novel nomogram model.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 disease patients confirmed by virus nucleic acid RT-PCR and CT

Exclusion Criteria:

* unconfirmed suspected cases
* Patients during pregnancy and lactation
* incomplete clinical data
* investigators considered patients ineligible for the trial
* Child patients

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: COVID-19 disease patients
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
the consistency of predicted severe rate and observed severe rate of COVID-19 patients | up to 3 months
  We aim to use the clinical data of COVID-19 patients to construct a nomogram model to predict the severe rate of each patient, then the the consistency of predicted severe rate and observed severe rate will be evaluated by calibration plot.
Duration of severe illness | up to 3 months
  the duration of severe illness of each patient will evaluated

CONTACTS AND LOCATIONS:
Locations (1):
- Xinqiao Hospital of Chongqing, Chongqing, Chongqing Municipality, China